CLINICAL TRIAL: NCT06213779
Title: A Multicentre, Prospective, Observational, 8-week Inception Cohort Study Being Carried Out by the Acute Respiratory Failure Section of China
Brief Title: The Burden of Acute Respiratory Failure in Chinese ICUs: a National Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, Professor, Southeast University, China
Other Study IDs: Chi-ARDS
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Acute Respiratory Failure; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- One group: This is a prospective observational study, aimed at collecting an adequate dataset on a large cohort of patients admitted to a large number of ICUs.

SUMMARY:
We aim to prospectively assess the burden, management and therapeutic approaches and outcomes of acute respiratory failure requiring respiratory support, during the winter months in China.

The purpose of this study is to provide new and current data on the disease burden of acute respiratory failure and ARDS. It will answer the following questions:

* The frequency and disease burden of acute respiratory failure in China;
* The incidence of ARDS based on the new global definition within this patient cohort.
* The mortality of ARDS within this cohort, and how does this vary based on ARDS categories and severity.
* The long-term outcomes (1-year mortality and survivor quality of life) of ARDS within this cohort.
* The nature course of ARDS (different stages and severity of ARDS).
* The respiratory support management strategies, such as recruitment maneuvers, prone positioning, ECCO2R, and ECMO.
* The use of drugs during ICU stays, including glucocorticoid, anticoagulant, nitric oxide, sivelestat, Xuebijing, and ulinastatin.
* The economical burden of acute respiratory failure within this patient cohort.
* The impact of occupation, incomes and education levels on the incidence and mortality of ARDS.

DETAILED DESCRIPTION:
1. The goal of this study will focus on the following items:

   * The frequency and disease burden of acute respiratory failure in China;
   * The incidence of ARDS based on the new global definition within this patient cohort.
   * The mortality of ARDS within this cohort, and how does this vary based on ARDS categories and severity.
   * The long-term outcomes (1-year mortality and survivor quality of life) of ARDS within this cohort.
   * The nature course of ARDS (different stages and severity of ARDS).
   * The respiratory support management strategies, such as recruitment maneuvers, prone positioning, ECCO2R, and ECMO.
   * The use of drugs during ICU stays, including glucocorticoid, anticoagulant, nitric oxide, sivelestat, Xuebijing, and ulinastatin.
   * The economical burden of acute respiratory failure within this patient cohort.
   * The impact of occupation, incomes and education levels on the incidence and mortality of ARDS.
2. Methods 2.1 Study Design This is a national prospective observational study, aimed at collecting an adequate dataset on a large cohort of patients admitted to a large number of ICUs in China. Each ICU will be requested to recruit for 8 consecutive 'winter' weeks between January 2024 and April 2024.

   2.2 Inclusion and exclusion criteria
   * Inclusion criteria: All patients admitted to the participating ICU receiving invasive, non-invasive ventilation or high-flow nasal cannula (HFNC) will be screened and included in the database.
   * Exclusion criteria:Age<18
3. Sample size calculation Our aim is to obtain a sample of at least 1500 ARDS patients within the cohort.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the participating ICU receiving invasive, non-invasive ventilation or high-flow nasal cannula (HFNC) will be screened and included in the database.

Exclusion Criteria:

* Age<18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our aim is to obtain a sample of at least 1500 ARDS patients within the cohort of patients receiving respiratory support.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Development of ARDS with new global definition | 28-days

SECONDARY OUTCOMES:
ICU mortality | 28-days

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - China-Japan friendship hospital, Beijin
  - Zhongda Hospital, Southeast university, Nanjing